CLINICAL TRIAL: NCT00885859
Title: Is Transcutaneous Electrical Nerve Stimulation (TENS) an Effective Method to Modulate Pain Transmission and Pain Perception in Patients Suffering From Chronic Non-Specific Pain Syndromes?
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) in Chronic Pain, Responders and Non-Responders?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: M. van Kleef, MaatrichtUMC
Other Study IDs: MEC 09-2-025
Record Dates: First submitted 2009-04-21; First posted 2009-04-22 (Estimated); Last update posted 2009-04-22 (Estimated); Status verified 2009-04

CONDITIONS: Neck Pain; Lower Back Pain; Shoulder Pain
MeSH Terms: conditions — Neck Pain; Low Back Pain; Shoulder Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: responders: patients who have a pain reduction of 30% or more after two weeks TENS-treatment
  Interventions: Device: TENStemeco Schwa Medico [Transcutaneous Electrical Nerve Stimulation (TENS)]
- 2: non-responders: patient who have a pain reduction smaller than 15% after two weeks TENS-treatment
  Interventions: Device: TENStemeco Schwa Medico [Transcutaneous Electrical Nerve Stimulation (TENS)]

INTERVENTIONS:
Device: TENStemeco Schwa Medico [Transcutaneous Electrical Nerve Stimulation (TENS)] — Patients are instructed how to use the TENS device during the two weeks at home.Self-adhesive reusable electrodes are used to deliver the electrical stimulation. The frequency is 100 Hz, pulse duration 250 μ sec. Stimulus intensity is strong but not unpleasant. The TENS electrodes are attached proximally and distally around the maximum pain point/area. Patients use TENS 4 times daily (30 minutes each time).
  Other Names: TENStemeco Schwa Medico

SUMMARY:
* Transcutaneous electrical nerve stimulation (TENS) is a frequently applied therapy in chronic pain. Although evidence regarding the effectiveness of TENS in chronic pain is inconclusive many patients continue using TENS on long term in daily practice. An important question is therefore why some patients respond well and others don't at all. In chronic pain evidence for abnormal pain processing (sensitization) has been found in several patients groups. The process of sensitization might influence effectiveness of TENS as the theoretical working mechanism of TENS is based on the modulation of the transmission of nociceptive impulses form peripheral receptors throughout spinal nerve system into the brain. In this study we want to study the effect of TENS on pain transmission, as measured by contact heat evoked potentials (CHEPS), between 'responders' and non-responders' after a two weeks TENS treatment. 'Responders' will be defined as patients with a pain reduction of ≥ 30% on a VAS after a two week treatment period with TENS. Non-responders are patients with a pain reduction < 15%.
* Objective: a) Is pain reducing effect TENS in responders based on modulation of pain transmission and perception, as measured by CHEPS? b) Is the ability of TENS to modulate pain transmission and perception influenced by abnormal pain processing?
* Prospective cohort study
* Patients with chronic non specific pain (duration > 6 months), above 18 year, will be included. Patients are referred from the Pain Clinic of the University Hospital Maastricht (MUMC). Exclusion criteria are: a) pain due to cancer, b) the use of a cardiac pacemaker, c) pregnancy, d) neurological sensory deficits, e) language and/or cognitive inability to complete the health assessment questionnaires f) previous TENS for pain relief.
* Patients receive a two week treatment period with TENS-treatment, as regular, at home after instruction. The frequency is set at 100 Hz and pulse duration at 250 μ sec. Patients have to use the TENS daily (minimal 4 times a day for 30 minutes).

Main study parameters/endpoints are decrease in amplitude of CHEPS in responders versus non-responders.

ELIGIBILITY:
Inclusion Criteria:

* referred for TENS treatment by a pain physician,
* duration of pain > 6 months,
* age above 18,
* no current other treatment for pain besides pain medication. Patients are allowed to continue their regular pain medication (as described by physician) prior to the TENS treatment

Exclusion Criteria:

* pain due to cancer,
* the use of a cardiac pacemaker,
* pregnancy,
* neurological sensory deficits,
* language and/or cognitive inability to complete the health assessment questionnaires
* previous TENS for pain relief.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic musculoskeltal pain will be recruted from the Pain Clinic of the University Hospital Maastricht (MUMC)
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2009-06; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Contact heat evoked potentials (CHEPS) | before and after two weeks treatment

SECONDARY OUTCOMES:
Severity of pijn on average past week(100mm VAS) | before and after two weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Kleef, Phd, MD, Study Director — Maastricht University Medical Center
Locations (1):
- MaastrichtUMC, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Buonocore M, Camuzzini N. Increase of the heat pain threshold during and after high-frequency transcutaneous peripheral nerve stimulation in a group of normal subjects. Eura Medicophys. 2007 Jun;43(2):155-60. Epub 2006 Oct 3. PMID 17021587
- [Background] de Tommaso M, Fiore P, Camporeale A, Guido M, Libro G, Losito L, Megna M, Puca F, Megna G. High and low frequency transcutaneous electrical nerve stimulation inhibits nociceptive responses induced by CO2 laser stimulation in humans. Neurosci Lett. 2003 May 15;342(1-2):17-20. doi: 10.1016/s0304-3940(03)00219-2. PMID 12727307
- [Background] de Tommaso M, Shevel E, Pecoraro C, Sardaro M, Divenere D, Di Fruscolo O, Lamberti P, Livrea P. Intra-oral orthosis vs amitriptyline in chronic tension-type headache: a clinical and laser evoked potentials study. Head Face Med. 2006 May 25;2:15. doi: 10.1186/1746-160X-2-15. PMID 16725028